CLINICAL TRIAL: NCT03185858
Title: System-integrated Technology-enabled Model of Care to Improve the Health of Stroke Patients in Rural China
Brief Title: SINEMA Model of Care to Improve the Health of Stroke Patients in Rural China
Acronym: SINEMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Collaborators: Medical Research Council (Other Government); Wellcome Trust (Other); Economic and Social Research Council, United Kingdom (Other); Department for International Development, United Kingdom (Other Government); Beijing Tiantan Hospital (Other); China Mobile Research Institute (Other); Xingtai Center for Disease Control and Prevention, China (Unknown); Centers for Disease Control and Prevention, China (Other Government); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015MRC0012
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: secondary prevention; primary healthcare; village doctors; rural China; medication adherence; physical activity
MeSH Terms: conditions — Stroke; Medication Adherence; Motor Activity

STUDY DESIGN:
Intervention Model Description: The SINEMA model, cognizant of health system's organization around primary, secondary and tertiary healthcare levels in China, adopts the principles of cascade training with feedback and task-sharing, and relies on existing human resources available at the community level. It also proposes the use of innovative mobile technology as tools (in the form of an Android-based SINEMA APP for village doctors and cellphone voice messages for participants). The overarching aim is to strengthen the capacity of village doctors on delivering services for the secondary prevention of stroke and promoting medication adherence and physical activity among stroke survivors.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors (staffs from a nearby county) are masked with no information on which villages will be assigned to intervention group or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SINEMA intervention group (Experimental): The intervention arm will implement the SINEMA model for one year, which consists of a provider-facing intervention aiming to strengthen the capacity of village doctors in delivering stroke secondary prevention, and a stroke survivor-facing intervention aiming to promote medication adherence and physical activity.
  Interventions: Behavioral: SINEMA intervention
- Control group (No Intervention): Villages in the control arm continue their usual practice without the introduction of any of the SINEMA activities described above. People who have hypertension or who are at high-risk of hypertension may receive follow-up visits four times per year as part of the basic public health services required by the government.

INTERVENTIONS:
Behavioral: SINEMA intervention — Provider-facing intervention includes the following components:
  (1) Systematic cascade training for village doctors; (2) monthly follow-up visits with the support of the SINEMA APP; (3) village doctor group activities; (4) performance feedback and incentives.
  Stroke survivor-facing intervention program includes the following components:
  (1) Briefing session; (2) monthly follow-up visits and follow-up handout; (3) daily voice message for health education.
  Arms: SINEMA intervention group

SUMMARY:
Despite the significant burden of stroke in rural China, secondary prevention of stroke is scarce. The aim of the study is to develop a system-integrated technology-enabled intervention (SINEMA) model for the secondary prevention of stroke in rural China and evaluate the effectiveness of the model compared with usual care. The hypothesis is that trained village doctors, equipped with digital health technology, can provide essential evidence-based care to stroke survivors in rural China.

DETAILED DESCRIPTION:
The SINEMA trial is a cluster-randomized controlled trial to evaluate the effectiveness of implementation of a system-integrated and technology-enabled model of care to improve the secondary prevention of stroke in Nanhe County, a rural area of Hebei province, China. Fifty villages from five townships are stratified randomized in a 1:1 ratio to either the intervention arm (implementing SINEMA model) or the control arm (usual care).

After a baseline survey, intervention will be implemented in 25 intervention villages, lasting for 12 months. Follow-up survey will be conducted in the same way in all villages at 12-month after the initial of the study. Process evaluation will be conducted every three month, and economic evaluation will also be conducted.

ELIGIBILITY:
Inclusion Criteria: those who

* are aged more than 18 years old;
* have a history of stroke (including ischemic and hemorrhagic stroke) diagnosed at county hospital or higher-level facilities, and currently in a clinically stable condition and not receiving acute stroke treatment;
* will live in this village for at least nine months during the next 12 months;
* have a basic communication ability (i.e. can understand simple instructions);
* give participant informed consent and are willing to participate in the study.

Exclusion Criteria: those who

* are unable to get out of bed without maximum assistance;
* have serious life-threatening disease such as cancers;
* who have an expected life span of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1299 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
systolic blood pressure | change from baseline to 12-month of follow-up
  change in systolic blood pressure

SECONDARY OUTCOMES:
mobility | change from baseline to 12-month of follow-up
  measured by timed-up-and-go test, a simple and quick functional mobility test that requires the participants to stand up, walk 3 meters, turn, walk back, and sit down
medication adherence | change from baseline to 12-month of follow-up
  measured using 4 item Morisky Green Levine Scale-4 (MMAS-4), which scores adherence from 0-4 and continuation of medication taking is measured by the total months of medication taking
physical activity level | change from baseline to 12-month of follow-up
  measured using the short version of the International Physical Activity Questionnaire(IPAQ)
health related quality of life | change from baseline to 12-month of follow-up
  measured using EuroQol-5 Dimensions-5L (EQ5D)
diastolic blood pressure | change from baseline to 12-month of follow-up
  participants' diastolic blood pressure

OTHER OUTCOMES:
stroke recurrence and hospitalization | at the end of the intervention (12-month)
  will be collected through questionnaire and medical insurance records
disability | at the end of the intervention (12-month)
  measured using modified Rankin Scale (ranged 0 (no symptom) to 5 severe disability)
Stroke related mortality | at the end of the intervention (12-month)
  will be collected through questionnaire, medical insurance records and verbal autopsy

CONTACTS AND LOCATIONS:
Overall Officials: Lijing L. Yan, PhD, Principal Investigator — Duke Kunshan Unviersity
Locations (1):
- Nanhe County, Xingtai, Hebei, China

IPD SHARING:
Plan to Share IPD: No
The investigators will not share the individual participant data. But other researchers could contact PI if there is special inquiry.

REFERENCES:
- [Derived] Yang B, Gong E, Chen X, Tan J, Peoples N, Li Y, Cai J, Li Y, Oldenburg B, Chen C, Dong D, Zhang X, Finkelstein E, Si L, Yan LL. Economic Evaluation of a Multicomponent mHealth Intervention for Stroke Management in Rural China: Cluster-Randomized Trial With 6-Year Follow-Up. JMIR Mhealth Uhealth. 2025 Sep 11;13:e75326. doi: 10.2196/75326. PMID 40934495
- [Derived] Gong E, Sun L, Long Q, Xu H, Gu W, Bettger JP, Tan J, Ma J, Jafar TH, Oldenburg B, Yan LL. The Implementation of a Primary Care-Based Integrated Mobile Health Intervention for Stroke Management in Rural China: Mixed-Methods Process Evaluation. Front Public Health. 2021 Nov 17;9:774907. doi: 10.3389/fpubh.2021.774907. eCollection 2021. PMID 34869187
- [Derived] Yan LL, Gong E, Gu W, Turner EL, Gallis JA, Zhou Y, Li Z, McCormack KE, Xu LQ, Bettger JP, Tang S, Wang Y, Oldenburg B. Effectiveness of a primary care-based integrated mobile health intervention for stroke management in rural China (SINEMA): A cluster-randomized controlled trial. PLoS Med. 2021 Apr 28;18(4):e1003582. doi: 10.1371/journal.pmed.1003582. eCollection 2021 Apr. PMID 33909607
- [Derived] Gong E, Yan LL, McCormack K, Gallis JA, Bettger JP, Turner EL. System-integrated technology-enabled model of care (SINEMA) to improve the health of stroke patients in rural China: Statistical analysis plan for a cluster-randomized controlled trial. Int J Stroke. 2020 Feb;15(2):226-230. doi: 10.1177/1747493019869707. Epub 2019 Aug 28. PMID 31462178
- [Derived] Wu N, Gong E, Wang B, Gu W, Ding N, Zhang Z, Chen M, Yan LL, Oldenburg B, Xu LQ. A Smart and Multifaceted Mobile Health System for Delivering Evidence-Based Secondary Prevention of Stroke in Rural China: Design, Development, and Feasibility Study. JMIR Mhealth Uhealth. 2019 Jul 19;7(7):e13503. doi: 10.2196/13503. PMID 31325288
- [Derived] Gong E, Gu W, Sun C, Turner EL, Zhou Y, Li Z, Bettger JP, Oldenburg B, Amaya-Burns A, Wang Y, Xu LQ, Yao J, Dong D, Xu Z, Li C, Hou M, Yan LL. System-integrated technology-enabled model of care to improve the health of stroke patients in rural China: protocol for SINEMA-a cluster-randomized controlled trial. Am Heart J. 2019 Jan;207:27-39. doi: 10.1016/j.ahj.2018.08.015. Epub 2018 Sep 5. PMID 30408621